CLINICAL TRIAL: NCT05800457
Title: The Role of Synovectomy in Pain Reduction Among Osteoarthritis Patients Following Total Knee Arthroplasty
Brief Title: The Role of Synovectomy in Pain Reduction Following Total Knee Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Brent Lanting, Orthopaedic Surgeon, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 12994
Record Dates: First submitted 2023-03-04; First posted 2023-04-05 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Total knee replacement with partial synovectomy (Experimental): Patients in this arm will undergo partial synovectomy during total knee replacement surgery.
  Interventions: Procedure: Partial synovectomy
- Total knee replacement without partial synovectomy (No Intervention): Patients in this arm will not undergo partial synovectomy during total knee replacement surgery.

INTERVENTIONS:
Procedure: Partial synovectomy — Patients in the intervention group will undergo partial synovectomy during total knee replacement surgery
  Arms: Total knee replacement with partial synovectomy

SUMMARY:
Osteoarthritis (OA) is the most common joint disease, causing severe pain due to joint inflammation (synovitis). While total knee arthroplasty (TKA) is commonly performed to reduce pain, 20% of patients are dissatisfied with their outcome post-surgery. This dissatisfaction is caused by persistent pain post-TKA due to synovitis that is not routinely removed during surgery. To address this problem, a synovectomy can be performed during TKA, which involves resecting the inflamed layer of tissue lining the joint, called the synovium, and its associated sensory nerve endings. Since the synovium will regenerate in the months post-surgery, synovectomy only transiently reduces pain after TKA. The proposed study will help ascertain the benefits and effects of synovectomy in patients who are more likely to experience poor satisfaction (driven mostly by pain) post-TKA. This study will include 62 patients undergoing TKA due to end-stage OA who have moderate to severe synovitis, as determined by ultrasound assessment. Patients will be randomized (1:1) to undergo a TKA with synovectomy or without synovectomy. Primary and secondary outcomes will be assessed through patient-reported levels of pain and function, results from physical performance tests, and quality of life (QOL) scores. These measures will be recorded pre- and post-surgery for comparison. Through demonstrating that synovectomy can at least transiently reduce pain post-TKA, this study will provide evidence for the development of medical therapies that target the synovium to slow its regrowth. This will be transformative for the long-term management of joint pain and synovitis post-surgery, thus significantly improving patients' overall QOL.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females over the age of 40 diagnosed with knee osteoarthritis
2. Scheduled for first unilateral total knee arthroplasty
3. Moderate to severe (at least grade two) synovitis and synovial hyperplasia, as determined by ultrasound assessment
4. Referred to the Pre-Admission Clinic at University Hospital

Exclusion Criteria:

1. Bilateral, uni-compartmental, or revision total knee arthroplasty
2. Osteoarthritis due to genetic syndromes (e.g., Ehlers-Danlos Syndrome, etc.)
3. Known inflammatory arthropathy, another rheumatic disease, or disease-modifying anti-rheumatic drug (DMARD) use (e.g. methotrexate, hydroxychloroquine, sulfasalazine, leflunomide, TNF inhibitors, etc.) - note: Gout is NOT an exclusion
4. Joint injection (steroid or viscosupplement) within 12 weeks of Pre-Admission Clinic appointment date
5. Cannot read, write, or understand English (printed instructions are provided in English only)
6. Any factors precluding patients from attending follow-up appointments (e.g., socio-economic limitations, distance from clinic, no access to home/cell phone, etc.).
7. Cognitive impairment or psychological problems that preclude the ability to understand instructions
8. Not able to follow up at routine standard of care post-operative visits

Ages: 41 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Patients' self-reported level of pain | 12 weeks post-surgery
  Pain will be measured using the pain sub-scale (nine items) of the Knee injury and Osteoarthritis Outcome Score (KOOS). Each question on the KOOS is a self-administered questionnaire is assigned a score from zero (no problems) to four (extreme problems) using a five-point Likert scale. The average of each sub-scale is calculated independently. Sub-scale scores range from zero (minimum), indicating severe knee problems, to 100 (maximum), indicating no knee problems (therefore, a higher score is better). The KOOS has demonstrated face validity and construct validity, as well as excellent test-retest reliability for each domain. It has also shown to be responsive to change in patients with knee OA.

SECONDARY OUTCOMES:
Joint function - 30-Second Sit to Stand Test | 6, 12, 18, and 24 weeks post-surgery
  The 30-Second Sit to Stand Test, which assesses leg strength and endurance in older adults, requires patients to complete as many full stands from the chair as possible in a 30-second time period. The number of full stands completed is compared to values that correspond to the patient's age group to determine their level of performance (a higher number is better).
Joint function - Timed Up and Go Test | 6, 12, 18, and 24 weeks post-surgery
  To begin the Timed Up and Go Test, patients will be seated in a chair. They will be signalled to stand up, walk to a line positioned three meters away from the chair, and walk back at a normal pace. Patients will then be instructed to return to their seated position. Patients' time, in seconds, will be recorded. Taking a longer time to perform this test indicates that the patient is less mobile, has a poorer sense of balance, and is at a higher risk of falling (taking a longer time is worse).
Patients' self-reported quality of life | 6, 12, 18, and 24 weeks post-surgery
  Quality of life will be evaluated using the European Quality of Life Five-Dimension (EQ-5D). The EQ-5D measures generic quality of life and consists of domains concluding mobility, self-care, usual activities, pain and discomfort, and anxiety and depression. Scores range from zero to one, with higher scores indicating a better quality of life. This tool has strong test re-test reliability and cross-sectional construct validity in patients with knee OA.
Symptoms sub-scale of the Knee injury and Osteoarthritis Outcome Score (KOOS) | 6, 12, 18, and 24 weeks post-surgery
  This sub-scale contains seven items. Each question on the KOOS self-administered questionnaire is assigned a score from zero (no problems) to four (extreme problems) using a five-point Likert scale. The average of each sub-scale is calculated independently. Sub-scale scores range from zero (minimum), indicating severe knee problems, to 100 (maximum), indicating no knee problems (therefore, a higher score is better). The KOOS has demonstrated face validity and construct validity, as well as excellent test-retest reliability for each domain. It has also shown to be responsive to change in patients with knee OA.
Activities of daily living sub-scale of the Knee injury and Osteoarthritis Outcome Score (KOOS) | 6, 12, 18, and 24 weeks post-surgery
  This sub-scale contains 17 items. Each question on the KOOS self-administered questionnaire is assigned a score from zero (no problems) to four (extreme problems) using a five-point Likert scale. The average of each sub-scale is calculated independently. Sub-scale scores range from zero (minimum), indicating severe knee problems, to 100 (maximum), indicating no knee problems (therefore, a higher score is better). The KOOS has demonstrated face validity and construct validity, as well as excellent test-retest reliability for each domain. It has also shown to be responsive to change in patients with knee OA.
Knee-related quality of life sub-scale of the Knee injury and Osteoarthritis Outcome Score (KOOS) | 6, 12, 18, and 24 weeks post-surgery
  This sub-scale contains four items. Each question on the KOOS self-administered questionnaire is assigned a score from zero (no problems) to four (extreme problems) using a five-point Likert scale. The average of each sub-scale is calculated independently. Sub-scale scores range from zero (minimum), indicating severe knee problems, to 100 (maximum), indicating no knee problems (therefore, a higher score is better). The KOOS has demonstrated face validity and construct validity, as well as excellent test-retest reliability for each domain. It has also shown to be responsive to change in patients with knee OA.
Inflammation | Ultrasound: Before surgery, 3 and 6 months post-surgery, Samples: Intra-operatively
  This will be measured through ultrasound scans pre- and post-surgery and by collecting synovial fluid and tissue samples intra-operatively.

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre - University Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No